CLINICAL TRIAL: NCT03741660
Title: Konjac-Mannan (Glucomannan) Improves Glycemia and Other Associated Risk Factors for Coronary Heart Disease in Type 2 Diabetes
Brief Title: Konjac-Mannan Improves Glycemia and Other Risk Factors for CHD in T2DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Dicofarm (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Konjac in T2DM
Record Dates: First submitted 2018-11-07; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Type2 Diabetes; Coronary Heart Disease
Keywords: konjac; type2 diabetes; fiber; coronary heart disease
MeSH Terms: conditions — Coronary Disease | interventions — (1-6)-alpha-glucomannan; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Konjac-mannan (Experimental): Konjac-mannan fiber-enriched biscuits with NCEP Step II metabolically controlled diet
  Interventions: Dietary Supplement: konjac glucomannan
- Placebo (Placebo Comparator): wheat bran fiber biscuits with NCEP Step II metabolically controlled diet
  Interventions: Dietary Supplement: wheat bran

INTERVENTIONS:
Dietary Supplement: konjac glucomannan — Konjac-mannan fiber-enriched biscuits (0.7 g/412KJ [100kcal] of glucommanan)
  Arms: Konjac-mannan
Dietary Supplement: wheat bran — Wheat bran (hard red wheat bran) fiber enriched biscuits
  Arms: Placebo

SUMMARY:
To examine whether Konjac-mannan fiber improves metabolic control measured by glycemia, lipidemia, and blood pressure in individuals with type-2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* hyperlipidemia controlled by medication
* hypertension controlled by medication
* type 2 diabetes controlled by medication
* minimum 3 years since onset of all three conditions
* sedentary lifestyle

Exclusion Criteria:

* regular smoking
* regular alcohol consumption
* family history of premature coronary heart disease
* hypothyroidism
* renal, hepatic or gastrointestinal disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1991-01 (Actual); Primary Completion 1992-06 (Actual); Study Completion 1998-06 (Actual)

PRIMARY OUTCOMES:
change in total:HDL cholesterol | change from baseline at week 3, relative to control
change in fructosamine | change from baseline at week 3, relative to control
change in systolic blood pressure | change from baseline at week 3, relative to control

SECONDARY OUTCOMES:
change in total cholesterol | change from baseline at week 3, relative to control
change in LDL cholesterol | change from baseline at week 3, relative to control
change in HDL cholesterol | change from baseline at week 3, relative to control
change in apolipoprotein A-1 | change from baseline at week 3, relative to control
change in apolipoprotain B | change from baseline at week 3, relative to control
change in glucose | change from baseline at week 3, relative to control
change in insulin | change from baseline at week 3, relative to control
diastolic blood pressure | change from baseline at week 3, relative to control
change in body weight | change from baseline at week 3, relative to control
change in apoB:ApoA-1 | change from baseline at week 3, relative to control